CLINICAL TRIAL: NCT06537258
Title: A Heart Rate Variability Biofeedback Enhanced Behavioral Intervention to Improve Psychological and Disease Functioning in Youth With Inflammatory Bowel Disease (IBD)
Brief Title: Heart Rate Variability and Inflammatory Bowel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Bonney Reed, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007611; R01DK139653-01 (NIH)
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Diseases
Keywords: cognitive behavioral therapy; heart rate variability
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback Enhanced Treatment (Experimental): Participants in this group will participate in biofeedback enhanced cognitive behaviorally based coping skills treatment. Treatment will consist of a 6-visit group intervention conducted online, via Emory zoom. Groups will include 5-8 patients. Groups will meet approximately each week for 6 weeks. Patients will also rate their disease symptoms and measures of clinical disease activity will be collected via chart review. Clinical assessments will occur at baseline within 1 week prior to starting treatment (T1), at treatment end or 6 weeks after baseline (T2), 14 weeks after baseline to capture 2-month follow-up after treatment (T3) and at 26 weeks after baseline (T4).
  Interventions: Behavioral: Biofeedback Enhanced Treatment
- Wait-list control (No Intervention): Participants randomized to the waitlist control group will complete the same assessment protocol at the time of randomization (Baseline) and again 6 weeks later. They will then be invited to begin treatment and will repeat the assessments at posttest and again at 14 and 26-week follow-up (for a total of 5 assessments).

INTERVENTIONS:
Behavioral: Biofeedback Enhanced Treatment — At all 4 assessment points (T1-T4), HRV will be measured using the ECG module of the mobile MindWare system at a sampling rate of 500 Hz, and a Skin Conductance Response (SCR) will be collected at a sampling rate of 10 Hz using eSense for iPad. Electrodes to assess SCR and HRV will be attached to patients during an ~10-minute period.
  A 5-minute initial baseline assessment will occur first followed by three 5-minute stress trials.
  Stress tasks will be audio recorded to measure study fidelity, and participants will be asked to rate their subjective level of stress with each trial. At all assessment points (T1-T4), participants will be provided with stool collection kits to collect a stool sample within 3 days of the laboratory psychophysiological assessment.
  At all assessment points (T1-T4), a blood draw of approximately 3 ml of blood will be collected.
  Other Names: biofeedback cognitive behaviorally based coping skills treatment
  Arms: Biofeedback Enhanced Treatment

SUMMARY:
The goals of this study are to test the effectiveness of a virtually delivered, group-based coping skills treatment program incorporating heart rate variability biofeedback to target autonomic dysfunction in youth diagnosed with inflammatory bowel disease (IBD). The investigators will enroll participants with IBD in a biofeedback enhanced cognitive behaviorally based coping skills treatment. Participants will be randomized to biofeedback enhanced treatment or wait-list control.

DETAILED DESCRIPTION:
The goals of this study are to test the effectiveness of a virtually delivered, group-based coping skills treatment program incorporating heart rate variability biofeedback to target autonomic dysfunction in youth diagnosed with inflammatory bowel disease (IBD).

Patients are youth ages 13-18 recruited through IBD clinics at Children's Healthcare of Atlanta. Enrollment will include up to 128 children with at least 1 parent. This study will last 7-months and will have 4 in person study visits, lasting about 1 hour each, as well as 6 virtual treatment sessions lasting about 45 minutes each.

Study procedures will include surveys, chart/record review, blood sampling, and non-invasive assessments of psychophysiological functioning. Stool samples will be collected and stored. Informed consent and assent will be obtained in-person or remote signed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with biopsy-confirmed IBD for at least 4 months,
* ages 13 through 18 years inclusive,
* speak English,
* enrolling with at least 1 parent/guardian who is willing to participate by completing surveys,
* positive depression or anxiety screens using the PHQ-4, - access to home internet to participate in virtual intervention,
* youth and parent agree to the conditions of study participation, including randomization, participation in intervention, and follow-up assessments,
* youth is medically approved to engage in normal daily activities (e.g., attend school, extracurricular activities)

Exclusion Criteria:

* previous diagnosis of developmental disabilities that require full-time special education or that impair the ability to respond to treatment,
* diagnosis with any other chronic disease (e.g., diabetes, epilepsy, etc.),
* diagnosis of abnormal thyroid function,
* treatment with any drug with known autonomic cardiovascular influences including beta-blockers, central sympatholytic agents, or antidepressants.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Changes in psychological distress | Baseline, 6 weeks post-intervention
  A continuous composite measure of stress, anxiety, and depression. Which will be analyzed continuously to evaluate for a significant mean difference between randomized groups at study endpoint (6-weeks). Scores range from 0 to 63, with higher scores indicating greater distress.

CONTACTS AND LOCATIONS:
Overall Officials: Bonney Reed, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Atlanta Metropolitan Area, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Center for Advanced Pediatrics, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with Researchers who provide a methodologically sound proposal. The research team will share individual participant data that underlie the results reported in a published article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 36 months following article publication.
Access Criteria: Proposals should be directed to ebreed@emory.edu To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website, Vivli.